CLINICAL TRIAL: NCT05887700
Title: A Multi-center, Single-arm, Real-world Registry Assessing the Clinical Use of the Lifetech CeraFlex™ ASD Closure System
Brief Title: Lifetech CeraFlex™ ASD Closure System Post-Market Clinical Follow-Up
Status: Recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT-TS-271-2023-01
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Atrial Septal Defect
Keywords: Lifetech; Atrial Septal Defect; ASD; CeraFlex; ASD Closure System
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ASD subjects: Patients with a confirmed diagnosis of Atrial Septal Defect (ASD) and implanted with the investigational device.
  Interventions: Device: CeraFlex™ Atrial Septal Defect (ASD) Closure System

INTERVENTIONS:
Device: CeraFlex™ Atrial Septal Defect (ASD) Closure System — The CeraFlex™ ASD Occluder have two types of occluders, CeraFlex™ ASD Occluder and CeraFlex™ Multi-fenestrated (Cribriform) ASD Occluder. The CeraFlex™ ASD Occluder is percutaneous, transcatheter closure devices for the non-surgical closure of atrial septal defects.

SUMMARY:
The objective of this post-market registry is to assess the clinical use of the Lifetech CeraFlex™ Closure System in a real-world and on-label fashion.

DETAILED DESCRIPTION:
The study intends to collect data from patients who have implanted with the device between 2019 and 2022. The data collection process is expected to complete by end of 2024. Final report shall be available in 2025.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of Atrial Septal Defect (ASD) and implanted with the investigational device as per IFU instructions.
2. Patients or legally authorized representatives have signed Data Release Consent or equivalent documents.

Exclusion Criteria:

Patients did not conduct any follow up visit after hospital discharge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of Atrial Septal Defect (ASD) and implanted with the investigational device.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 6 months post-implantation
  Procedural success is defined as a composite of:
  1. Absence of stroke/TIA, device embolization, cardiac or vascular perforation or device/procedure related death, assessed at 6 months post-implantation.
  2. Successful closure of the defects, with no, trivial or small residual shunt confirmed by Doppler echocardiography at 6 months post-implantation.

SECONDARY OUTCOMES:
Incidence of moderate or large residual shunt | At procedure, 6 months and 12 months post-implantation
Incidence of device or procedure related Adverse Events (AEs) | From attempted procedure to 24 months post-implantation
Incidence of device or procedure related Serious Adverse Events (SAEs) | From attempted procedure to 24 months post-implantation
Incidence of Device Deficiencies (DD) | From attempted procedure to 24 months post-implantation
Incidence of death | From attempted procedure to 24 months post-implantation

CONTACTS AND LOCATIONS:
Locations (7):
- Brazil (5):
  - Hospital Pequeno Príncipe, Curitiba
  - Universidade Federal do Ceará, Fortaleza
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - HCOR - Associação Beneficente Síria, São Paulo
  - Hospital Beneficência Portuguesa, São Paulo
- Onassis Cardiac Surgery Center, Kallithea, Greece
- IRCCS Policlinico San Donato, Milan, Italy

IPD SHARING:
Plan to Share IPD: No